CLINICAL TRIAL: NCT01565356
Title: Comparison of PET Images Acquired at 30 Min and 50 Min Post Injection of 18F-AV-45 in Healthy Volunteers and Alzheimer's Disease Patients
Brief Title: Evaluation of PET Scan Timing Relative to AV-45 Injection Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A06
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer's Disease
Keywords: Amyloid imaging; Positron Emission Tomography; 18F-AV-45; florbetapir F 18; Diagnostic imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: florbetapir F 18 — IV injection, 111 or 370MBq (3 or 10mCi), single dose
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
This study will re-read 10-minute positron emission tomography (PET) scans acquired in previous clinical studies of AV-45 at 30 and 50 minutes after injection and compare the results.

ELIGIBILITY:
Eligibility for subjects scans to be used in this study is determined by subject's eligibility/enrollment in Study A01(NCT01565291) or A03(NCT01565330).

Inclusion Criteria (AD group):

* Greater than 50 years of age
* Probable AD according to the National Institute of Neurological and Communication Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* Mild/moderate dementia as evidenced by a Mini-Mental State Examination (MMSE) score ranging from 10 to 24, boundaries included, at screening
* History of cognitive decline gradual in onset and progressive over a period of at least 6 months

Inclusion Criteria (A01[NCT01565291] healthy volunteer group):

* 50 years of age, inclusive

  * MMSE of 29 or greater

Inclusion Criteria (A03[NCT01565330] healthy volunteer group):

* 35 to 55 years of age, inclusive
* MMSE of 29 or greater

Exclusion Criteria (both groups):

* Neurodegenerative disorders other than AD, including, but not limited to Parkinson's disease, Pick's disease, fronto-temporal dementia, Huntington's chorea, Down syndrome, Creutzfeldt-Jacob disease, normal pressure hydrocephalus, and progressive supranuclear palsy
* Diagnosis of other dementing / neurodegenerative disease
* Diagnosis of mixed dementia
* Cognitive impairment resulting from trauma, hypoxic damage, vitamin deficiency, brain infection, brain cancer, endocrine disease, or mental retardation
* Clinically significant infarct or possible multi-infarct dementia as defined by the NINCDS criteria
* Evidence on screening MRI or other biomarker that suggests alternate etiology for cognitive deficit (for healthy controls, evidence suggesting the presence of AD pathology)
* Clinically significant psychiatric disease
* History of epilepsy or convulsions
* Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances
* Current clinically significant cardiovascular disease
* Received investigational medication within the last 30 days

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NO SUBJECTS WERE ENROLLED IN THIS STUDY - this study re-read scans obtained in other clinical studies
Groups:
- All Subject Scans: 22 florbetapir-PET scans obtained in Study A01 and and 19 scans obtained in A03
Period: Overall Study
Arm/Group | All Subject Scans
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Subject Scans
Number analyzed (Participants) | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 65.49 (15.302)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Percent Agreement of Interpretation Between 30-40 and 50-60 Min Reads - Qualitative Evaluation
Description: Three independent readers blinded to subject identification, subject diagnosis, subject demographics and PET scan time points post-injection read each scan and reported as amyloid positive or amyloid negative. Results show the percentage of agreement between the majority read of 30-40 min scan and the majority read of the 50-60 min scan.
Time Frame: Scans acquired 30-40 min and 50-60 min after injection
Measure: Number; unit: percentage of agreement
Groups:
- All Scans: 22 florbetapir-PET scans obtained in Study A01(NCT01565291) and and 19 scans obtained in A03(NCT01565330)
Arm/Group | All Scans
Number analyzed (Participants) | 41
percentage of agreement | 100
Statistical Analysis 1: Comparison: All Scans; Cohen's (simple) kappa statistic; Test type: Superiority or Other; Kappa statistic = 1.00, 95% CI 2-sided [1.00 to 1.00]

2. Secondary Outcome: Agreement of Interpretation Between 30-40 and 50-60 Min Reads - Semi-quantitative Evaluation
Description: Three independent readers blinded to subject identification, subject diagnosis, subject demographics and PET scan time points post-injection read each scan and reported the results using a 5-point scale (0=no amyloid; 4=high levels of amyloid deposition). Results are reported as a weighted kappa statistic.
Time Frame: Scans acquired 30-40 min and 50-60 min post-injection
Measure: Number (95% Confidence Interval); unit: weighted kappa
Arm/Group | All Scans
Number analyzed (Participants) | 41
weighted kappa | 0.946 [0.906 to 0.987]

ADVERSE EVENTS:
Description: No subjects received florbetapir in this study. This study consisted of rereads of scans previously acquired in other clinical studies (A01,A03).
Arm/Group | All Subject Scans
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days